CLINICAL TRIAL: NCT06342323
Title: Study on the Optimal Number of Fiducial Marker Implanted With 3D-template Assitance for Stereotactic Body Radiotherapy
Brief Title: The Optimal Number of Fiducial Marker for Stereotactic Body Radiotherapy
Acronym: ONFM-SBRT
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Qiu Bin, Doctor-in-charge, Peking University Third Hospital
Other Study IDs: IRB00006761-M2023235; ONFM-SBRT (Other: Peking university third hospital)
Record Dates: First submitted 2024-03-19; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer; Liver Cancer; Pancreatic Cancer; Renal Cell Carcinoma
Keywords: fiducial marker; SBRT; lung caner; liver cancer; pancreatic cancer; renal cell carcinoma
MeSH Terms: conditions — Lung Neoplasms; Liver Neoplasms; Pancreatic Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fiducial marker group: all patient is observed for SBRT treatment error after fiducial marker implantation.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — the fiducial marker was implanted with 3D template assistance under CT guidance

SUMMARY:
This is a clinical study focused on the use of fiducial marker-guided stereotactic body radiotherapy (SBRT) for treating malignant tumors, including lung, liver, pancreatic, and kidney/adrenal cancers. Here's a breakdown of the key components of the study:

Study Design: Prospective, single-center, exploratory clinical study.

Patient Enrollment: The study intends to enroll patients diagnosed with malignant tumors requiring fiducial marker-guided SBRT. Each tumor type (lung, liver, pancreatic, kidney/adrenal) aims to include 15 cases.

Informed Consent: Patients are required to sign informed consent before participating in the study, indicating their understanding of the procedures, risks, and benefits involved.

Intervention: Enrolled patients will undergo stereotactic radiotherapy for their respective malignant tumors. During this process, fiducial markers will be implanted according to the study protocol.

Monitoring: Following implantation of fiducial markers, the study will monitor adverse events associated with the procedure. This includes any complications or side effects resulting from the marker implantation process.

Success Rate: The study will assess the success rate of fiducial marker implantation. This likely involves evaluating the accuracy and reliability of marker placement for guiding SBRT treatment.

SBRT Treatment Error: The study will also monitor SBRT treatment errors. This involves tracking any deviations or inaccuracies in the delivery of stereotactic radiotherapy, potentially caused by issues such as improper fiducial marker placement or technical errors in treatment administration.

Overall, the study aims to explore the feasibility and effectiveness of using fiducial marker-guided SBRT for treating various types of malignant tumors to assess both the safety and the efficacy with a focus on patient outcomes and treatment accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with lung cancer, liver cancer, renal cancer, pancreatic cancer.
* Going to have SBRT.

Exclusion Criteria:

* Needle insertion route impeded by skeletal structures and close to blood vessels which have high risks of puncture bleeding;
* Poor organ function (e.g. poorly controlled high blood pressure);
* Poor compliance, unable to complete coordination;
* Participant who is considered inappropriate or unwilling to participate in this clinical trial for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with lung cancer, liver cancer, renal cancer, pancreatic cancer who going to have fiducial marker guided SBRT was all eligible.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2023-10-08 (Actual); Primary Completion 2024-10-07 (Estimated); Study Completion 2025-10-07 (Estimated)

PRIMARY OUTCOMES:
success rate | 3 months after fiducial marker implantation during the SBRT
  the success rate of SBRT

SECONDARY OUTCOMES:
Treatment error | 3 months after fiducial marker implantation during the SBRT
  Error in fiducial marker tracking during each fraction of SBRT

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kothary N, Heit JJ, Louie JD, Kuo WT, Loo BW Jr, Koong A, Chang DT, Hovsepian D, Sze DY, Hofmann LV. Safety and efficacy of percutaneous fiducial marker implantation for image-guided radiation therapy. J Vasc Interv Radiol. 2009 Feb;20(2):235-9. doi: 10.1016/j.jvir.2008.09.026. Epub 2008 Nov 18. PMID 19019700